CLINICAL TRIAL: NCT02484326
Title: Development and Validation of a Clinical Risk Score Predicting the Cardiac Rupture in Patients With ST-elevation Myocardial Infarction
Brief Title: Clinical Risk Score Predicting the Cardiac Rupture in Patients With ST-elevation Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, MD, Chinese PLA General Hospital
Other Study IDs: 14FCJJ01
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-05

CONDITIONS: Cardiac Rupture
Keywords: ST-elevation myocardial infarction; Cardiac rupture; Risk assessment
MeSH Terms: conditions — Heart Rupture; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Grouping by different risk stratification — A simple risk score system based on 7 baseline clinical variables divided patients into four groups
  Other Names: Risk stratification

SUMMARY:
The purpose of this study is to validate a practical risk score to predict the mechanical complication of ST-elevation myocardial infarction (STEMI).

DETAILED DESCRIPTION:
STEMI patients chewed 300 mg aspirin and 600 mg clopidogrel in the emergency department, followed by oral 100 mg aspirin and 75mg clopidogrel daily for at least 12 months. STEMI patients received low molecular weight heparin (LMWH), β-blockers, and angiotensin converting enzyme inhibitors (ACEI) or angiotensin receptor blockers (ARB) according to the STEMI guideline, unless there were contraindications to these drugs. Peripheral blood samples were collected from patients within 2 hours of admission for blood routines and blood biochemistry examinations. White blood cell counts and level of hemoglobin were assessed with automated cell counters via standard techniques. The investigators followed up patients in validation group for three month to observe the cardiac rupture events and other adverse cardiac events .

ELIGIBILITY:
Inclusion Criteria:

ST-elevation myocardial infarction: concurrence of symptoms (chest pain or symptoms compatible with acute heart failure or unexplained syncope) and electrocardiogram findings (new onset left bundle branch block or ST-segment elevation≥1 mm in ≥2 inferior leads or ≥2 mm in ≥2 precordial leads)

Exclusion Criteria:

cancer mental illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ST-elevation myocardial infarction patients who were admitted from January 2012 to January 2013
Sampling Method: Non-Probability Sample
Enrollment: 3779 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiac rupture | 3 month
  Pericardial tamponade or electromechanical dissociation accompanied with massive pericardial effusion is the indicator of cardiac rupture

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Pouleur AC, Barkoudah E, Uno H, Skali H, Finn PV, Zelenkofske SL, Belenkov YN, Mareev V, Velazquez EJ, Rouleau JL, Maggioni AP, Kober L, Califf RM, McMurray JJ, Pfeffer MA, Solomon SD; VALIANT Investigators. Pathogenesis of sudden unexpected death in a clinical trial of patients with myocardial infarction and left ventricular dysfunction, heart failure, or both. Circulation. 2010 Aug 10;122(6):597-602. doi: 10.1161/CIRCULATIONAHA.110.940619. Epub 2010 Jul 26. PMID 20660803
- [Result] French JK, Hellkamp AS, Armstrong PW, Cohen E, Kleiman NS, O'Connor CM, Holmes DR, Hochman JS, Granger CB, Mahaffey KW. Mechanical complications after percutaneous coronary intervention in ST-elevation myocardial infarction (from APEX-AMI). Am J Cardiol. 2010 Jan 1;105(1):59-63. doi: 10.1016/j.amjcard.2009.08.653. PMID 20102891
- [Result] Figueras J, Barrabes JA, Serra V, Cortadellas J, Lidon RM, Carrizo A, Garcia-Dorado D. Hospital outcome of moderate to severe pericardial effusion complicating ST-elevation acute myocardial infarction. Circulation. 2010 Nov 9;122(19):1902-9. doi: 10.1161/CIRCULATIONAHA.109.934968. Epub 2010 Oct 25. PMID 20975001
- [Result] Lopez-Sendon J, Gurfinkel EP, Lopez de Sa E, Agnelli G, Gore JM, Steg PG, Eagle KA, Cantador JR, Fitzgerald G, Granger CB; Global Registry of Acute Coronary Events (GRACE) Investigators. Factors related to heart rupture in acute coronary syndromes in the Global Registry of Acute Coronary Events. Eur Heart J. 2010 Jun;31(12):1449-56. doi: 10.1093/eurheartj/ehq061. Epub 2010 Mar 15. PMID 20231153
- [Result] Jones BM, Kapadia SR, Smedira NG, Robich M, Tuzcu EM, Menon V, Krishnaswamy A. Ventricular septal rupture complicating acute myocardial infarction: a contemporary review. Eur Heart J. 2014 Aug 14;35(31):2060-8. doi: 10.1093/eurheartj/ehu248. Epub 2014 Jun 26. PMID 24970335
- [Result] Qian G, Liu HB, Wang JW, Wu C, Chen YD. Risk of cardiac rupture after acute myocardial infarction is related to a risk of hemorrhage. J Zhejiang Univ Sci B. 2013 Aug;14(8):736-42. doi: 10.1631/jzus.B1200306. PMID 23897793
- [Result] Roberts WC, Burks KH, Ko JM, Filardo G, Guileyardo JM. Commonalities of cardiac rupture (left ventricular free wall or ventricular septum or papillary muscle) during acute myocardial infarction secondary to atherosclerotic coronary artery disease. Am J Cardiol. 2015 Jan 1;115(1):125-40. doi: 10.1016/j.amjcard.2014.10.004. Epub 2014 Oct 13. PMID 25456862
- [Derived] Qian G, Jin RJ, Fu ZH, Yang YQ, Su HL, Dong W, Guo J, Jing J, Guo YL, Chen YD. Development and validation of clinical risk score to predict the cardiac rupture in patients with STEMI. Am J Emerg Med. 2017 Apr;35(4):589-593. doi: 10.1016/j.ajem.2016.12.033. Epub 2016 Dec 15. PMID 28132793